CLINICAL TRIAL: NCT01543022
Title: First in Man Study - a Prospective, Multicenter, Single Arm Trial to Investigate the Safety and Feasibility of the Symphony Device
Brief Title: Symphony: The Implantable Counter Pulsation Device (CPD) Safety and Feasibility Trial
Acronym: Symphony
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 184916
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Symphony system (Experimental)
  Interventions: Device: Symphony; Procedure: The operative approach is limited to an infraclavicular incision similar to that used for placement of a pacemaker

INTERVENTIONS:
Device: Symphony — The Symphony system has been developed for superficial implantation without the need to enter the chest. It allows for complete patient mobility and provides counter pulsation therapy for up to 30 days in hospitalized patients.
Procedure: The operative approach is limited to an infraclavicular incision similar to that used for placement of a pacemaker — The vascular graft is surgically attached (anastomosed) to the subclavian artery. The symphony device is implanted into a pocket below the pectoralis muscle on the anterior chest and attached to the graft. The driveline is tunneled out through the skin and attached to the drive console.

SUMMARY:
The Counter Pulsation Device (CPD) System 'Symphony' is intended to provide counter pulsation therapy for up to thirty (30) days to patients with chronic heart failure who have persistent worsening of their condition despite optimal medical therapy. Patients will be in New York Heart Association (NYHA) Class IIIb or IV heart failure and have exhausted all medical or surgical options.

ELIGIBILITY:
Inclusion Criteria:

1. New York Heart Association Class IIIB or IV heart failure despite optimal medical therapy, including ACE inhibitors, beta blockers, IV diuretics and pressors
2. Left Ventricular Ejection Fraction < 40%.
3. Patient is not a candidate for conventional catheter-based or surgical intervention such as valve intervention or coronary artery bypass surgery.
4. Patient is not currently a candidate for heart transplantation or placement of a left ventricular assist device (LVAD) as bridge to heart transplantation due to co-morbidities. Patients may become a candidate for these options if they have improvement on the device due to improved cardiac output.
5. Patients have exhausted all approved surgical and medical therapies as determined by a heart failure cardiologist and a surgeon with expertise in heart failure.
6. Patient has been evaluated by a multi-disciplinary research team and felt to be a suitable candidate for a research study. The final decision regarding the patient's candidacy for research will remain with the attending cardiologist and heart surgeon.
7. Improved hemodynamics on device support will allow for potential for physical rehabilitation.
8. Signed Informed Consent, or oral informed consent with written confirmation by uninvolved third party
9. Age of subject at least 19 years

Exclusion Criteria:

1. High likelihood of death during the current hospitalization (as judged by the attending physician) and condition other than heart failure that would limit survival to less than two years.
2. Require mechanical ventilation.
3. Failure to wean from IABP, Impella, ECMO or other mode of circulatory support.
4. Complex arrhythmias that negatively impact the effectiveness of counter pulsation.
5. Dependency on high dose inotropes.
6. Cerebrovascular accident or TIA within the previous 3 months.
7. Contraindication to anticoagulation medication such as Heparin, Coumadin, Aspirin and Plavix.
8. Presence of hypercoaguable state or history of idiopathic venous or arterial thrombosis.
9. Severe calcification in the target vessel that will preclude insertion of the Symphony device.
10. Moderate to severe aortic insufficiency (2+ or more).
11. Ongoing systemic infection defined as two of the following:

    * WBC > 12,500
    * positive blood culture
    * fever
12. Abnormal pre-albumin (< 13mg/dL), or albumin (< 3.0 mg/dl)
13. A cardiac rhythm that cannot be used to trigger the CPD (sinus rhythm, ventricular or atrial pacing, A-V pacing).
14. Abnormal bilateral carotid Doppler or CT exam define as > 50% stenosis.
15. Subclavian artery internal diameter of < 7 mm on Doppler study or CT exam.
16. Ability to ambulate < 200 metres on a 6 minute walk test.
17. Any aortic aneurysmal disease.
18. Active documented HIT.
19. Presence of mechanical heart valve.
20. Moderate to severe RV failure.
21. Severe tricuspid regurgitation.
22. History of major psychiatric illness.
23. End-organ dysfunction including:

    * renal failure defined as serum Cr > 2.5 mg/dl,
    * liver dysfunction defined as bilirubin 2X normal, or elevated INR with no anticoagulation,
    * respiratory failure defined as FEV1 < 50% predicted.
24. Chest X-ray to rule out pulmonary pathology that increases the risk of need for treatment prior to device implant.
25. BMI > 40 kg/ m2.
26. Active participation in another clinical trial that may interfere with this trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Death, Stroke or Transient Ischemic Attack (TIA), Limb Ischemia requiring surgical intervention | hospital discharge or 30 days of support, whichever is longer
  The trial will primarily look at patient safety defined as proportion of composite Major Adverse Events (MAE) up to hospital discharge or 30 days of CPD support, whichever is longer.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences Center, University Hospital, London, Ontario
  - Royal Victoria Hospital, Montreal, Quebec